CLINICAL TRIAL: NCT05395104
Title: A Phase 1, Open-label, 1-sequence Crossover, Drug-drug Interaction Study to Assess the Effect of Repeated Doses of Cefiderocol on the Pharmacokinetics of Midazolam in Healthy Adult Participants
Brief Title: A Study to Assess the Effect of Cefiderocol on the Pharmacokinetics (PK) of Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2136R2118
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Midazolam; Cefiderocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cefiderocol Plus Midazolam (Experimental): A total of 2 doses of midazolam and 45 doses of cefiderocol was administered to each participant per specified dosing schedule.
  Interventions: Drug: Midazolam; Drug: Cefiderocol

INTERVENTIONS:
Drug: Midazolam — Syrup for oral administration
Drug: Cefiderocol — Liquid for intravenous infusion

SUMMARY:
The purpose of this study is to determine the effect of repeated doses of cefiderocol on the PK of midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation, including medical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead electrocardiography at the Screening Visit and upon admission to the clinical research unit (CRU).
* Body weight ≥ 50 kilograms (kg) and body mass index within the range of ≥ 18.5 to ≤ 32.0 kg/meter squared at the Screening Visit.

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Systolic blood pressure outside the range of 90 to 145 millimeters of mercury (mmHg), diastolic blood pressure outside the range of 50 to 95 mmHg, pulse rate outside the range of 40 to 100 beats per minute, or blood pressure or pulse values considered clinically significant by the investigator at the Screening Visit or upon admission to the CRU. Abnormal values may be retested once.
* Lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Past use of over-the-counter or prescription medication, including herbal medications, traditional Chinese medicines, vitamins, minerals, dietary supplements, and vaccines within 14 days (or 5 terminal half-lives, whichever is longer) prior to admission to the CRU (which will occur on Day -2) or intended use of any of the above throughout the study enrollment.
* Significant blood loss of ≥ 500 milliliters or blood or plasma donation within 56 days prior to the Screening Visit until completion of the study, or from the Screening Period until admission to the CRU through completion of the study.
* History of coronavirus disease 2019 (COVID-19) infection within 14 days prior to the Screening Visit or admission, or close contact with a COVID-19 patient in the days prior to the Screening Visit or admission as reported by the participant and the participant's medical history.
* History of drug or alcohol abuse/addiction.
* Regularly consumes excessive amounts of caffeine, defined as > 6 servings of coffee, tea, caffeinated soft drinks, or other caffeinated beverages per day (1 serving is approximately equivalent to 120 milligrams of caffeine).
* Used tobacco- or nicotine-containing products (including cigarette, pipe, cigar, chewing tobacco, nicotine patch, or nicotine gum) within 6 months prior to admission to the CRU or refuses to refrain from using tobacco- or nicotine-containing products throughout the study (including Follow-up Period).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefiderocol Plus Midazolam: A total of 2 doses (5 milligrams [mg] each) of midazolam and 45 doses (2 grams [g] each) of cefiderocol were administered to each participant per specified dosing schedule.
Period: Overall Study
Arm/Group | Cefiderocol Plus Midazolam
Started | 14
Received At Least 1 Dose Of Study Drug (Safety Analysis Population) | 14
Completed | 12
Not Completed | 2
Not completed — Met Liver Stopping Criteria | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population: all participants who were exposed to study intervention.
Groups:
- Cefiderocol Plus Midazolam: A total of 2 doses (5 mg each) of midazolam and 45 doses (2 g each) of cefiderocol were administered to each participant per specified dosing schedule.
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. Cmax is reported as nanograms/milliliter (ng/mL). Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: Pharmacokinetics Parameter Population: All participants with at least 1 pharmacokinetics parameter estimated appropriately. Participants in the "Midazolam + Cefiderocol" population with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
ng/mL
  Midazolam Alone | 25.3 (45.3)
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 28.8 (35.0)
Statistical Analysis 1: Comparison: Cefiderocol Plus Midazolam; Midazolam + Cefiderocol: single 5-mg dose of midazolam + 2 g cefiderocol (Day 15); Test type: Other — Ratio = Geometric least squares mean (test)/geometric least squares mean (reference); Ratio = 1.0865, 90% CI 2-sided [0.9724 to 1.2141]

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. Tmax is reported in hours (hrs). Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: as for outcome 1
Measure: Median (Full Range); unit: hrs
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
hrs
  Midazolam Alone | 0.51 [0.50 to 1.00]
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 0.51 [0.50 to 1.07]

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. AUC0-last was calculated using the linear up/log down trapezoidal method and is reported as nanograms times hours/milliliter (ng*hrs/mL). Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hrs/mL
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
ng*hrs/mL
  Midazolam Alone | 66.13 (46.3)
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 77.37 (44.2)
Statistical Analysis 1: Comparison: Cefiderocol Plus Midazolam; Midazolam + Cefiderocol: single 5-mg dose of midazolam + 2 g cefiderocol (Day 15); Test type: Other — Ratio = Geometric least squares mean (test)/geometric least squares mean (reference); Ratio = 1.1174, 90% CI 2-sided [0.9784 to 1.2762]

4. Primary Outcome: Area Under the Concentration-time Curve Extrapolated From Time 0 to Infinity (AUC0-inf) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. AUC0-inf was calculated as: AUC0-last + [Clast/λz], where Clast is the last measured concentration and λz is the plasma terminal elimination rate constant on Days -1 and 15. Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hrs/mL
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
ng*hrs/mL
  Midazolam Alone | 68.69 (47.8)
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 81.07 (45.6)
Statistical Analysis 1: Comparison: Cefiderocol Plus Midazolam; Midazolam + Cefiderocol: single 5-mg dose of midazolam + 2 g cefiderocol (Day 15); Test type: Other — Ratio = Geometric least squares mean (test)/geometric least squares mean (reference); Ratio = 1.1239, 90% CI 2-sided [0.9887 to 1.2776]

5. Primary Outcome: Terminal Elimination Half-life (t1/2,z) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. t1/2,z was calculated as: (ln2)/λz on Days -1 and 15. Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hrs
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
hrs
  Midazolam Alone | 5.39 (33.7)
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 6.10 (41.7)

6. Primary Outcome: Terminal Elimination Rate Constant (λz) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. λz is the magnitude of the slope of the linear regression of the log concentration versus time profile during the terminal phase on Days -1 and 15 and is reported as 1/hours (1/h). Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hrs
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
1/hrs
  Midazolam Alone | 0.1287 (33.7)
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 0.1135 (41.7)

7. Primary Outcome: Mean Residence Time (MRT) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. MRT was calculated as: AUMC0-inf/AUC0-inf, and AUMC0-inf is the area under the first moment curve extrapolated to infinity on Days -1 and 15. Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hrs
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
hrs
  Midazolam Alone | 4.86 (26.5)
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 5.51 (33.4)

8. Primary Outcome: Apparent Total Clearance (CL/F) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. CL/F was calculated as: Dose/AUC0-inf on Days -1 and 15 and is reported as liters/hr. Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hr
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
liters/hr
  Midazolam Alone | 69.3 (60.3)
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 61.7 (45.6)

9. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Midazolam
Description: This outcome measure presents the effects of repeated doses of cefiderocol on the pharmacokinetics of midazolam. Vz/F was calculated as: Dose/AUC0-inf/λz on Days -1 and 15 and is reported as liters. Day -1 is defined as Baseline.
Time Frame: 0 (predose) up to 24 hours postdose on Day -1 (Midazolam alone at Baseline) and Day 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 14
liters
  Midazolam Alone | 538 (38.4)
  Midazolam + Cefiderocol: number analyzed (Participants) | 12
  Midazolam + Cefiderocol | 543 (52.2)

10. Secondary Outcome: Cmax of Cefiderocol
Description: This outcome measure presents the pharmacokinetics of cefiderocol when coadministered with midazolam. Cmax is reported as micrograms/milliliter (μg/mL).
Time Frame: Day 15
Population: Pharmacokinetics Parameter Population: All participants with at least 1 pharmacokinetics parameter estimated appropriately. Participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 11
μg/mL | 80.5 (21.8)

11. Secondary Outcome: Tmax of Cefiderocol
Description: This outcome measure presents the pharmacokinetics of cefiderocol when coadministered with midazolam.
Time Frame: Day 15
Population: as for outcome 10
Measure: Median (Full Range); unit: hrs
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 11
hrs | 2.92 [2.90 to 2.98]

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Dosing Interval τ (8 Hours) (AUC0-τ) of Cefiderocol
Description: This outcome measure presents the pharmacokinetics of cefiderocol when coadministered with midazolam. AUC0-τ was calculated by the linear up/log down trapezoidal method and is reported as micrograms times hours/milliliter (μg*hrs/mL).
Time Frame: Day 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hrs/mL
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 11
μg*hrs/mL | 355.4 (20.2)

13. Secondary Outcome: CL of Cefiderocol
Description: This outcome measure presents the PK of cefiderocol when coadministered with midazolam. CL was calculated as: Dose/AUC0-τ on Day 15.
Time Frame: Day 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hr
Arm/Group | Cefiderocol Plus Midazolam
Number analyzed (Participants) | 11
liter/hr | 5.63 (20.2)

ADVERSE EVENTS:
Time Frame: Day -1 through Day 23
Groups:
- Cefiderocol Plus Midazolam: A total of 2 doses of midazolam and 45 doses of cefiderocol were administered to each participant per specified dosing schedule.
Arm/Group | Cefiderocol Plus Midazolam
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cefiderocol Plus Midazolam (N=14)
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Infusion site extravasation (General disorders) | 7
Infusion site pain (General disorders) | 4
Infusion site phlebitis (General disorders) | 4
Catheter site pain (General disorders) | 2
Chills (General disorders) | 1
Infusion site dermatitis (General disorders) | 1
Infusion site inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Vessel puncture site haemorrhage (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1/9 — This adverse event only affected female participants..
Blood lactate dehydrogenase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT05395104/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT05395104/SAP_001.pdf